CLINICAL TRIAL: NCT03057275
Title: Performance of the Monica Novii Wireless Patch System in Pre-term Labor
Status: Completed | Type: Observational
Sponsor: GE Healthcare (Industry)
Responsible Party: Sponsor
Other Study IDs: 107-CT-007rev10_UAMC
Record Dates: First submitted 2017-02-15; First posted 2017-02-20 (Actual); Last update posted 2021-02-09 (Actual); Status verified 2021-02

CONDITIONS: Premature Labor
Keywords: Threatened Premature Labor; Abdominal Fetal ECG
MeSH Terms: conditions — Obstetric Labor, Premature

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

GROUPS / COHORTS (2):
- Threatened PTL: abdominal fetal/maternal monitoring
  Interventions: Device: Abdominal fetal/maternal monitoring
- Delivered PTL: abdominal fetal/maternal monitoring
  Interventions: Device: Abdominal fetal/maternal monitoring

INTERVENTIONS:
Device: Abdominal fetal/maternal monitoring — A single patch placed on the abdomen that incorporates 5 electrodes and a monitoring device
  Other Names: Novii Wireless Patch System

SUMMARY:
To study the equivalence of the Monica Novii™ Patch System in patients admitted for threatened pre-term labor and for pre-term labor & delivery from 32 +0 weeks gestation by determining the equivalence of the Novii™ Patch System in monitoring Fetal Heart Rate (FHR), Maternal Heart Rate (MHR) and Uterine Contractions (UC) to Doppler FHR, tocodynamometer (TOCO) UC and photo plethysmograph MHR FDA approved predicates.

DETAILED DESCRIPTION:
The study is a single-center prospective paired comparison trial, to determine the equivalence of the Monica Novii Patch System with FDA cleared Doppler FHR, TOCO UC and photo plethysmograph MHR Predicate. Patients admitted for threatened pre-term labor and for pre-term labour & delivery will be monitored with both devices simultaneously for FHR, UC, and MHR. Only the data from predicate devices will be available to the clinical care team. The equivalence of the Novii data will be compared to that of the simultaneously obtained predicate device data.

Since TOCO UC and Doppler FHR are prone to artefact or error in a Pre-Term Labor population, the principal investigator or a member of the study team will decide on:

1. One 30 minute period of 'interpretable' Doppler FHR, photo plethysmograph MHR and TOCO UA from each of the admitted threatened pre-term labor subjects, when the subject is experiencing contractions as demonstrated by the TOCO UC trace and these contractions represent the clinical presentation.
2. One 30 minute period of 'interpretable' Doppler FHR, photo plethysmograph MHR and TOCO UA from each of the pre-term labor & delivery subjects ending as close to delivery as practical. As above the TOCO UC contractions should represent the clinical presentation.

The selection of the 30 min periods will be based on data from the predicate only (the Novii FHR and UC data will not be available to the study team).

The two 30 min periods will be used for the statistical equivalence calculation. All recorded data will be made available for visual review.

ELIGIBILITY:
Inclusion Criteria:

* She will require pre-term labor (at least 32 weeks 0 days gestation) monitoring with a singleton longitudinal, breech, transverse lie pregnancy.
* She had none of the exclusion criteria.

Exclusion Criteria:

The presence of any of the following factors or conditions would exclude the patient from consideration as a subject:

* Known major fetal malformation or chromosome abnormality.
* Multiple gestation
* A condition for which cesarean will likely be carried out shortly.
* Involvement in another clinical trial currently or previously in this pregnancy that, in the investigator's opinion, would affect the conduct of this study.
* Medical or obstetric problem that would preclude the use of abdominal electrodes (e.g., skin eruptions, history of sensitivity to adhesives).
* Parturient is under age 18.
* Medical or obstetric problem that in investigator's opinion would make the patient incapable of taking part in the study.
* Inability to understand the consent information due to medical illness or diminished intellectual capacity, or insurmountable language barrier.
* Potential for coercion, e.g. Prisoners.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subjects admitted for threatened pre-term labor (total of 30 subjects) will be recruited for the study according to the following strata:
  * 15 patients with a gestation equal to 32 weeks +0 days gestation but < 34 weeks +4 days
  * 5 patients with a Body Mass Index (BMI) less than 29
  * 5 patients with a BMI equal to 29 but less than 35
  * 5 patients with a BMI equal to or more than 35
  * 15 patients with a gestation equal to 34 weeks +4 days gestation but < 37 weeks +0 days
  * 5 patients with a BMI less than 29
  * 5 patients with a BMI equal to 29 but less than 35
  * 5 patients with a BMI equal to or more than 35
  Subjects admitted for pre-term labor & delivery (total of 30 subjects) will be recruited for the study following the same stratification plan as above.
Sampling Method: Non-Probability Sample
Enrollment: 47 (Actual)
Dates: Start 2017-04-20 (Actual); Primary Completion 2019-09-20 (Actual); Study Completion 2019-09-20 (Actual)

PRIMARY OUTCOMES:
FHR Percent Agreement | 30min
  The fetal heart rate output file from the predicate device is processed to generate a time line plot of FHR data in which the epochs with un-interpretable data (e.g. no FHR value in that 2 second window) are removed to create "interpretable" only FHR data, i.e. the predicate is represented as 100% successful. A corresponding Monica Novii file is then generated that has the same time epochs as the Doppler FHR data set but containing the Novii FHR data or uninterpretable data (i.e. no FHR value).
FHR Bland Altman | 30min
  Bland-Altman plots will be provided separately for each subject, together with an overall assessment using all available data from all subjects. For this overall assessment, the hierarchical nature of the dataset will be taken into account in the statistical analysis. An appropriate statistical approach is described by Bland and Altman , although in practice the analysis may also be accomplished by using a mixed model method.
FHR Deming Regression | 30min
  Standard linear regression of y on x is not appropriate in this situation as the predicate device is not considered a gold standard, but as a device providing a measurement which may itself be subject to error, whereas the standard linear regression method assumes x to be measured without error. Deming regression is a method for calculating the regression line y=α+βx when both variables are subject to error, and the ratio of the error variances in x and y is known (and will be assumed to be equal to 1 in this analysis).
UC percent agreement | 30min
  The positive percentage agreement (PA) is determined separately for each subject from the interpretable and uninterpretable data as follows:
  PA (%)=(a/(a+C))×100 Equation 3
  Where:
  "a" is the number of minutes when both the Monica Novii Pod/Patch and the predicate devices are "interpretable" at the same time "c" is the number of minutes when the Predicate is "interpretable" but the Monica Novii Pod/Patch is "un-interpretable".
  This can be alternatively described as using only those times when the Predicate device gives "Interpretable" data, and is defined as the percentage of those times for which the Monica Novii Pod/Patch also gives "Interpretable" data (i.e. it is analogous to sensitivity but based on reliability).
UC Positive percent agreement | 30min
  The Positive Percent Agreement PPA of the Novii System against the Predicate will be determined from the "individual contraction "detection as follows:
  PPA(%)=(x/(x+z))×100 Equation 4
  Where:
  "x" is the total number of "individual contractions" detected by BOTH the Novii Pod/PATCH and the Predicate "z" is the total number of "individual contractions" detected by the Predicate only.
  Again the test for statistical non-inferiority of percent agreement based on individual uterine contractions will be defined as in Equation 2 for a one-sided 95% confidence interval using t=1.70.
MHR percent agreement | 30min
  As for FHR
MHR bland altman | 30min
  As for FHR
MHR deming regression | 30min
  As for FHR

CONTACTS AND LOCATIONS:
Overall Officials: Megahan G Hill, MBBS, Principal Investigator — Banner- University of Arizona Medical Center
Locations (1):
- University of Arizona Medical Center, Tucson, Arizona, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Gonzalez M, Hill M, Cohen WR. Performance of a Maternal Abdominal Surface Electrode System for Fetal Heart Rate and Uterine Contraction Monitoring from 34 to 37 Weeks. Am J Perinatol. 2024 Feb;41(3):263-269. doi: 10.1055/a-1673-1765. Epub 2021 Oct 19. PMID 34666382